CLINICAL TRIAL: NCT02036151
Title: Impact of Maternal Xylitol Consumption on Mutans Sterptococci ,Plaque and Caries Levels in Children
Brief Title: Impact of Maternal Xylitol Consumption on Mutans Sterptococci
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Najlaa Alamoudi, Prof. Chairman Preventive Dental Sciences, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KAU
Record Dates: First submitted 2013-12-31; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Dental Caries and Streptococcus Mutans Count
Keywords: Xylitol; prevention; Mutans streptococci; caries; plaque; children
MeSH Terms: conditions — Dental Caries; Plaque, Amyloid | interventions — Xylitol; Chewing Gum; Tablets; sodium fluoride topical preparation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental, control (Experimental): Mothers in the experimental group were instructed to chew 1 pellet of xylitol gum (Fennobon Oy, Yrittäjäntie, Finneland -gum, 3 times ) for a period of 3 months. control mothers did not receive any medications. All mothers received oral hygiene instructions and restorative treatment when needed. Offspring of both the experimental and control groups did not receive any medication and were followed for at 6,12, 18 and 24 month from initiation of mothers consumption. month
  Interventions: Drug: xylitol
- fluoride varnish application (Active Comparator): The control group participated in a preventive program under the supervision of the Pediatric Dentistry Department. The program activities consisted of oral hygiene instructions, fluoride varnish application (Duraphat 5% Na F ,Ultradent Products, Utah, USA) and restorative treatment when needed.
  Interventions: Drug: fluoride varnish application

INTERVENTIONS:
Drug: xylitol — Mothers in the experimental group were instructed to chew 1 pellet of xylitol gum (Fennobon Oy, Yrittäjäntie, Finneland -gum, 3 times ) for a period of 3 months. control mothers did not receive any medications. All mothers received oral hygiene instructions and restorative treatment when needed. Offspring of both the experimental and control groups did not receive any medication and were followed for at 6,12, 18 and 24 month from initiation of mothers consumption. month
  Other Names: Fennobon Oy, Yrittäjäntie, Finneland - chewing; gum, tablet , 1.8g and containing 66% xylitol by weight,
  Arms: Experimental, control
Drug: fluoride varnish application — The control group participated in a preventive program under the supervision of the Pediatric Dentistry Department. The program activities consisted of oral hygiene instructions, fluoride varnish application (Duraphat 5% Na F ,Ultradent Products, Utah, USA) and restorative treatment when needed.
  Other Names: fluoride varnish (Duraphat 5% Na F ,Ultradent Products, Utah, USA)
  Arms: fluoride varnish application

SUMMARY:
The study was designed to determine whether maternal xylitol consumption through regular chewing of xylitol gums can affect the salivary mutans streptococci (MS), dental caries, and dental plaque levels of their children.

DETAILED DESCRIPTION:
Method: Study sample included 60 mother and child pairs with high salivary mutans streptococcus (MS) levels. Samples were randomly divided into experimental group (30 pairs) and control group (30 pairs). Mothers in the experimental group received xylitol chewing gum treatment three times/day for three months, whereas the controls received fluoride varnish. Both groups received oral hygiene instructions, dietary counseling and restorative treatment. All children were examined after 6, 12 and 18 months from the initiation of the study to assess caries, plaque and salivary mutans streptococcus (MS) levels.

ELIGIBILITY:
Inclusion Criteria:

* mothers with high salivary counts (≥ 105)
* mothers having children at least 10 months of age (10-36months) or having a minimal of 8 primary teeth.

Exclusion Criteria:

* subjects with systemic disorders or on regular medications

Ages: 10 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Assesment of mutans streptococci count in off-spring | 24 month
  Collection of saliva samples was carried out for microbiological screening after 6, 12, 18 and 24 months from the initiation xylitol consumption .Un stimulated saliva samples were collected from each child for salivary bacterial level screening. Saliva sampling was performed before conducting the clinical examination between 9-11 am. Children were not allowed to eat or drink for 2 hours before sampling. Saliva was collected with the pipette supplied by the dentocult (CRT) kit. (Ivoclar Vivadent, Lichtenstein). Saliva sample was not taken if the child has received antibiotics within 1 month prior the examination. Screening of stimulated saliva samples for mutans streptococcus (MS) level were carried out using the dentocult method (CRT). Findings of 105 CFU or more of MS indicates a high caries risk, whereas findings less than 105 CFU is considered low caries risk.

SECONDARY OUTCOMES:
Assesment of Caries level in off-spring | 24 month
  Clinical examination was carried out for dmft score for deciduous teeth after 6, 12, 18 and 24 months from the initiation maternal xylitol consumption. The diagnosis of dental caries was based on the WHO criteria 1987.
  .

CONTACTS AND LOCATIONS:
Locations (1):
- King abulaziz University, Dental University Hospital, Jeddah, P.O Box 80209, Saudi Arabia

REFERENCES:
- [Result] Alamoudi NM, Hanno AG, Sabbagh HJ, Masoud MI, Almushayt AS, El Derwi DA. Impact of maternal xylitol consumption on mutans streptococci, plaque and caries levels in children. J Clin Pediatr Dent. 2012 Winter;37(2):163-6. doi: 10.17796/jcpd.37.2.261782tq73k4414x. PMID 23534323